CLINICAL TRIAL: NCT06012500
Title: Evaluation of Explanted Lungs by MRI and Biological Assays
Acronym: Xe MRI in ILD
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0031
Record Dates: First submitted 2021-09-03; First posted 2023-08-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: ILD
MeSH Terms: interventions — Xenon-129

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy Controls
  Interventions: Drug: Xenon-129
- ILD: Participants with diagnosed ILD
  Interventions: Drug: Xenon-129

INTERVENTIONS:
Drug: Xenon-129 — Inhaled contrast for MRI

SUMMARY:
The purpose of this multi-centered, NIH-sponsored study is to to develop an optimal protocol for using non-invasive 129Xe gas exchange MRI to detect changing disease activity in interstitial lung diseases (ILDs). We base this study on the demonstrated promise of 129Xe as a biomarker for both prognosis and therapy response, overwhelming interest from both industry and academic partners, and impending FDA approval for 129Xe ventilation MRI. This requires disseminating standardized and repeatable methods for 3D 129Xe functional MRI in order to facilitate innovative multi-center observational and interventional trials that can advance our understanding of fibrotic lung disease, while accelerating the development of novel therapies.

DETAILED DESCRIPTION:
There remains an urgent need to better phenotype interstitial lung diseases, predict trajectories, monitor progression, and measure treatment response. Because ILD pathology is spatially and temporarly heterogeneous, the problem demands a 3-dimensional (3D) lung assessment. To this end, CT imaging patterns are critical in IPF diagnosis, but such structural imaging is insensitive to changing functional status. Thus, we have developed hyperpolarized (HP) 129Xe MRI, whose unique properties enable rapid, non-invasive, 3D functional assessment of inhaled gas distribu-tion in the airspaces, as well as its uptake in the pulmonary interstitium (barrier tissues) and trans-fer to the pulmonary capillary red blood cells (RBCs). This way of probing regional gas exchange confers sensitivity to micron-scale interstitial barrier thickening and locally diminished RBC trans-fer. We have used 129Xe MRI to predict outcomes such as death or the need for transplant and have provided preliminary evidence showing that barrier uptake is a sensitive and early marker of therapy response. These advancements have led to demands for wider dissemination, which drives an urgent need to harmonize acquisition protocols and quantification methods.

This work will be conducted by 4 collaborating centers - Duke University, the University of Cin-cinnati, Cincinnati Children's Hospital Medical Center, and the University of Wisconsin. Cincin-nati Children's will operate under its own IRB protocol and IND, but each will share data and im-aging techniques in order to establish best practices. The specific aims of the work are:

Aim 1 - Maximize and Measure Repeatability of 129Xe MRI/MRS Metrics across MRI Platforms. We will improve upon published repeatability of ±15-20% by harmonizing MRI/MRS protocols by improved coaching, optimized dose delivery, and tailoring the inhaled dose volume to the individ-ual patient. Using these approaches, each center will demonstrate coefficients of repeatability of ±6% or better in patients with ILD.

Aim 2 - Establish Harmonized Quantitative Analysis of Gas Exchange MRI/MRS. We will deploy a reconstruction and analysis package enabling users of any of three major MRI vendor plat-forms to obtain robust, real-time quantitative analysis of images and spectra. We will demon-strate that healthy reference cohorts are equivalent to ±10% across 4 centers and use this to build the definitive multi-site healthy reference distributions.

Aim 3 - Deploy a Clinical Framework to Identify Active Fibrosis and Normal Aging. To position the technology for clinical deployment and interpretation, we will develop a physiologic model incorporating ventilation, barrier and RBC metrics to explain the underlying factors responsible for a given patient's diffusing capacity (DLCO) and transfer coefficient (KCO). This framework will be deployed to readers who will differentiate ILD from normal aging.

The expected outcomes are to 1) deploy robust and standardized acquisition and analysis proto-cols across centers and scanner platforms, 2) establish the methods and standards for maximiz-ing repeatability of each gas exchange imaging metric, and 3) provide the tools and framework needed to use 129Xe MRI to characterize disease and assess therapeutic efficacy. Collectively, this program will enable rapid and innovative trials that will accelerate progress in studying and treating fibrotic lung disease. While this technical development study is focused on healthy sub-jects and those with ILD, deployment of these non-invasive MRI methods should benefit the study of interstitial lung disease more broadly, as well as other conditions of gas exchange im-pairment such as pulmonary vascular disease, COPD, and COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients of either gender, age > 18
2. Willing and able to give informed consent and adhere to visit/protocol schedules (Consent must be given before any study procedures are performed.)
3. Clinical diagnosis of Interstitial Lung Disease made by a board certified pulmonologist us-ing established criteria. We will not exclude individuals based on ILD type or severity of disease with the exception of the below criteria

Exclusion Criteria:

1. Subject is less than 18 years old
2. MRI is contraindicated based on responses to MRI screening questionnaire
3. Subject is pregnant or lactating
4. Resting oxygen saturation on room air <90%
5. Respiratory illness of a bacterial or viral etiology within 30 days of MRI
6. Subject has history of any known ventricular cardiac arrhythmia
7. Subject has history of cardiac arrest within the last year
8. Subject does not fit into 129Xe vest coil used for MRI
9. Subject cannot hold his/her breath for 15 seconds
10. Subject deemed unlikely to be able to comply with instructions during imaging
11. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Patients with ILD and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximize and Measure Repeatability of 129Xe MRI/MRS Metrics across MRI Platforms | 1 day
  Harmonize MRI/MRS protocols by improved coaching, optimized dose delivery, and tailoring the inhaled dose volume to the individual patient. Using these approaches, each center will demonstrate coefficients of repeatability of ±6% or better in patients with ILD.
Establish Harmonized Quantitative Analysis of Gas Exchange MRI/MRS | 1 day
  Deploy a reconstruction and analysis package enabling users of any of three major MRI vendor platforms to obtain robust, real-time quantitative analysis of images and spectra.
Deploy a Clinical Framework to Identify Active Fibrosis and Normal Aging | 1 Day
  To position the technology for clinical deployment and interpretation, we will develop a physiologic model incorporating ventilation, barrier and RBC metrics to explain the underlying factors responsible for a given patient's diffusing capacity (DLCO) and transfer coefficient (KCO)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woods, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No